CLINICAL TRIAL: NCT00696293
Title: Optimizing Outcomes in Older Adults With Low Back Pain and Depression
Brief Title: Duloxetine Treatment of Major Depression and Chronic Low Back Pain For Older Adults
Acronym: ACHIEVE2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Jordan F. Karp, Associate professor, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KL2RR024154 (NIH)
Record Dates: First submitted 2008-06-09; First posted 2008-06-12 (Estimated); Results first posted 2016-05-26 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Major Depressive Disorder; Back Pain; Aged
MeSH Terms: conditions — Depressive Disorder, Major; Back Pain | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Duloxetine + clinical management
  NOTE -- THIS WORK WAS CONDUCTED AS PART OF A CAREER DEVELOPMENT AWARD. THE CLINICALTRIALS.GOV DESCRIPTION OF THE STUDY WAS UPDATED 1/5/16 TO UPDATE THE OPEN LABEL NATURE OF THIS WORK. THIS IS WHAT IS REPORTED HERE AND HAS BEEN PEER REVIEWED AND PUBLISHED.
  Interventions: Drug: Duloxetine

INTERVENTIONS:
Drug: Duloxetine — Duloxetine up to 120 mg/day + Clinical Management
  Other Names: Duloxetine = Cymbalta

SUMMARY:
The following primary hypotheses will be tested:

1. During Step 1: Major Depressive Disorder (MDD) or Chronic Low Back Pain (CLBP) in < 40% of the initial 60 subjects treated with duloxetine (DUL) + Clinical Management(CM) during the first 8 weeks will respond (response is defined as a Montgomery Asberg Depression Rating Scale (MADRS) score </=9 and at least a 30% improvement in back pain as measured with the 20-point numeric rating scale.
2. During Step 2: More DUL+Problem Solving Therapy for Depression and Pain (PST-DP) than DUL+CM treated subjects will achieve response during the second 8 weeks, defined as a MADRS score </=9 and at least a 30% improvement in back pain as measured with the 2-point numeric rating scale.
3. Improvement in depression scores will be correlated with improvement in CLBP scores.

The exploratory hypotheses to be tested are that:

During Step 2: Compared to subjects treated with DUL+CM, subjects treated with DUL+PST-DP will have improved outcomes in: 1) disability, 2) sleep, 2) functioning/quality of life, 3) caregiver burden/depression, and 5) analgesic use.

DETAILED DESCRIPTION:
This is a two-part study. Step 1 is an 8-week long open-label trial of duloxetine (DUL) + clinical management (CM), titrated up to 90 mg/day, for older adults with comorbid major depressive disorder (MDD) and chronic low back pain (CLBP). At week 8, if subjects have not responded, the dose of duloxetine is increased to 120 mg/day. Duloxetine will be increased and continued at 120 mg/day (or highest tolerated dose) for both randomized study groups (during step 2) to assure medication parity.

Step two starts at week 9 and includes those subjects whose MDD and/or CLBP has not met criteria for response during Step 1. At week 9 subjects will be randomized to receive treatment with either: 1) DUL 120 mg/day (or the highest tolerated dose)+ Problem Solving for Depression and Pain (PST-DP) or 2) DUL 120 mg/day (or highest tolerated dose) + CM. Step 2 will be delivered over the course of 8-10 sessions.

NOTE ADDED 1/5/16: THIS WAS TREATMENT DEVELOPMENT WORK CONDUCTED AS PART OF A CAREER DEVELOPMENT AWARD. ONLY THE FIRST OPEN-LABEL PART OF THE STUDY WAS COMPLETED, AND THESE RESULTS HAVE BEEN PUBLISHED AND WILL BE REPORTED HERE ON CLINICALTRIALS.GOV

ELIGIBILITY:
Inclusion Criteria:

* Age >/= 60
* Current episode of MDD per SCID DSM-IV criteria
* Must score >/= 16 on the CES-D assessment
* Serum sodium >/=130 mEq/ml
* CLBP of at least moderate severity for more days than not for >/= 3 months
* MADRS score >/= 15
* Sufficiently medically stable to be able to participate in a depression treatment protocol
* Willingness and ability to speak English Access to translators is limited. It would be unsafe to treat an older adult who does not speak English with an antidepressant and not be able to effectively communicate with them about their progress and any side effects. We provide a 24/7 on-call service for all subjects enrolled in this study. The on-call clinicians and physicians are not bilingual, and if a problem arose, it may be impossible to effectively interpret and manage the emergent situation. Finally, many of the assessments used in the study are self-reports. At the present time, we do not have the ability to translate these instruments into other languages. If the subject cannot read and understand English, this would interfere with their ability to complete the self-report assessments
* Willingness to discontinue other antidepressants and anxiolytics, except for lorazepam up to 2 mg/day
* Mini Mental State Exam > 20
* Willingness to provide informed consent
* Corrected visual ability that enables reading of newspaper headlines and hearing capacity that is adequate to respond to a raised conversational voice.

Exclusion Criteria:

* Meet DSM-IV criteria for dementia
* History of bipolar, schizophrenia, schizoaffective, or other psychotic disorder
* Alcohol or other drug abuse (including abuse of prescription medications) within the past 6 months
* History of treatment non-adherence in other protocols run by the Mid-Life or Late-Life Centers
* Acute pain superimposed on chronic pain. For example, subjects who report "red flags" which suggest a herniated disk, vertebral fracture, infection, cauda equina syndrome, or other medical emergency will be excluded
* Wheelchair bound
* History of documented non-response to duloxetine
* Concurrent use of thioridazine
* Active suicidal ideation with plan
* Uncontrolled narrow angle glaucoma

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-05; Primary Completion 2010-03 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jordan F Karp, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh School of Medicine, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Karp JF, Weiner DK, Dew MA, Begley A, Miller MD, Reynolds CF 3rd. Duloxetine and care management treatment of older adults with comorbid major depressive disorder and chronic low back pain: results of an open-label pilot study. Int J Geriatr Psychiatry. 2010 Jun;25(6):633-42. doi: 10.1002/gps.2386. PMID 19750557

RESULTS

PARTICIPANT FLOW:
Groups:
- Duloxetine Plus Clinical Management: Duloxetine + clinical management
  Duloxetine: Duloxetine up to 120 mg/day + Clinical Management
Period: Overall Study
Arm/Group | Duloxetine Plus Clinical Management
Started | 30
Completed | 28
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Duloxetine Plus Clinical Management
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.4 (7.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 9

OUTCOME MEASURES:

1. Primary Outcome: Change in Montgomery Asberg Depression Rating Scale(MADRS) Score From Baseline and 12 Weeks
Description: The MADRS is a rating of depression severity with theoretical scale range 0-60, with lower values representing better outcome
  Larger reduction between MADRS from baseline to 12 weeks would represent better outcome
Time Frame: baseline and 12 weeks
Population: description of median change
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine Plus Clinical Management
Number analyzed (Participants) | 28
units on a scale | -11.7 (6.5)

2. Primary Outcome: Change in McGill Pain Questionaire, Short Form, Score From Baseline and 12 Weeks
Description: The McGill Pain Questionaire, short form consists of 15 descriptors (11 sensory; 4 affective) which are rated on an intensity scale as 0 = none, 1 = mild, 2 = moderate or 3 = severe. The McGill Pain Questionaire score ranged from 0 (none) to 45 (severe).
  A larger reduction of the score from baseline to 12 weeks would represent a better outcome
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Duloxetine + Clinical Management: Duloxetine + clinical management
  NOTE -- THIS WORK WAS CONDUCTED AS PART OF A CAREER DEVELOPMENT AWARD. THE CLINICALTRIALS.GOV DESCRIPTION OF THE STUDY WAS UPDATED 1/5/16 TO UPDATE THE OPEN LABEL NATURE OF THIS WORK. THIS IS WHAT IS REPORTED HERE AND HAS BEEN PEER REVIEWED AND PUBLISHED.
  Duloxetine: Duloxetine up to 120 mg/day + Clinical Management
Arm/Group | Duloxetine + Clinical Management
Number analyzed (Participants) | 28
units on a scale | -6.0 (1.9)

ADVERSE EVENTS:
Arm/Group | Duloxetine Plus Clinical Management
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No